CLINICAL TRIAL: NCT05403489
Title: Comparison of the Results of Bronchoalveolar Lavage Culture and Endotracheal Aspirate Culture in Intubated Critically Ill COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Basri Cakiroglu (Other)
Responsible Party: Sponsor-Investigator, Basri Cakiroglu, Hisar Intercontinental Hospital, Hisar Intercontinental Hospital
Organization: Hisar Intercontinental Hospital (Other)
Other Study IDs: HisarIH
Record Dates: First submitted 2022-06-02; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Bronchoalveolar Lavage; COVID-19 Pneumonia; Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group B (bronchoalveolar lavage): Patients who underwent BAL* were named Group B
  * BAL: bronchoalveolar lavage
  Interventions: Procedure: Bronchoalveolar lavage
- Group E (endotracheal aspirate): Patients who received ETA** were named Group E.
  ** ETA: Endotracheal aspirate
  Interventions: Procedure: endotracheal aspirate culture

INTERVENTIONS:
Procedure: Bronchoalveolar lavage — In cases approved for bronchoscopy, bronchoalveolar lavage was performed and culture analysis was performed.
  Other Names: Bronchoalveolar lavage culture; fiberoptic bronchoscopy
  Groups: Group B (bronchoalveolar lavage)
Procedure: endotracheal aspirate culture — In cases where consent for bronchoscopy could not be obtained, tracheal secretions were aspirated and culture analysis was performed.
  Groups: Group E (endotracheal aspirate)

SUMMARY:
Introduction: Secondary pneumonia is frequently seen in COVID-19 cases followed up intubated, and high mortality rates can be observed. Isolation of the agent with bronchoalveolar lavage (BAL) culture or endotracheal aspirate (ETA) culture may increase the success of treatment. This study aimed to retrospectively analyze the results of BAL and ETA cultures in intubated COVID-19 cases.

Methods: We routinely apply BAL culture with bronchoscopy or ETA culture within the first 48 hours after intubating. We retrospectively screened cases who underwent BAL and ETA. They were divided into two groups: Group B and E. Evaluated parameters were compared in both groups.

Results: Demographic data and blood test results were similar in both groups. Intensive care unit (ICU) and intubation durations, and culture positivity were statistically significantly higher in Group B. Although not statistically significant, the mortality rate was higher in Group E. The most growth microorganisms were Candida species.

Conclusion: Mortality rates were consistent with the literature. Since the microorganism isolation rate is higher with BAL and antimicrobial treatment is applied more effectively; early deaths were prevented and stay periods were prolonged. In contrast, these durations were shorter in the ETA group due to higher mortality. In intubated COVID-19 cases, a more effective treatment process can be carried out by clearing the airway with fiberoptic bronchoscopy and by specifically planning the treatment according to the BAL culture. This may have a positive effect on prognosis and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Intubated COVID-19 patients
* Above 18 years old patients

Exclusion Criteria:

* Non COVID-19 patients
* Non intubated COVID-19 patients
* Below 18 years old patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who were intubated due to COVID 19 in our reanimation unit between January 2021 and December 2021 and underwent BAL or ETA analysis were retrospectively scanned from the hospital information management system and patient files.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Culture positivity | 1 years
  Significantly higher microbiological culture growth rate was obtained in Group B
Length of stay in intensive care unit | 1 years
  Significantly higher duration of stay in intensive care unit was found in Group B
Duration of intubation | 1 years
  Significantly higher duration of stay intubated was observed in Group B
Mortality | 1 years
  Mortality rate was higher in Group E. But not statistically significant.

SECONDARY OUTCOMES:
Microorganism | 1 years
  The most growing microorganism in both groups was the Candida species.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Huseyin Kilic, Principal Investigator — Hisar Intercontinental Hospital
Locations (1):
- Hisar Intercontinental Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No